CLINICAL TRIAL: NCT01735266
Title: Comparative Efficacy of Whole-colon Water Exchange, Left-colon Water Exchange and Air Methods of Colonoscopy on Cecum Intubation in Unsedated Outpatients - - - a Prospective, Randomized Controlled Trail
Brief Title: Left-colon WEC May Reduce Insertion Time Compared With Whole-colon WEC.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 20121108-5
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Polyp; Pain
Keywords: Colonoscopy
MeSH Terms: conditions — Polyps; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Air colonoscopy (Active Comparator): Air was insufflated during whole procedure of colonoscope insertion.
  Interventions: Other: Air colonoscopy
- Whole-colon water exchange colonoscopy (Experimental): The air pump was turned off before colonoscopy. During the whole procedure of the scope insertion, residual air in lumen was suctioned and 37°C (maintained with a water bath) water was infused with a peristaltic pump to obtain lumen visualization. Air was insufflated until cecum was reached or appendix opening was seen.
  Interventions: Other: Water exchange colonoscopy
- left-colon water exchange colonoscopy (Experimental): In the left side of colon (including descending colon, sigmoid colon and rectum), water was infused instead of air to obtain lumen visualization as described above in whole-colon water exchange colonoscopy group.
  Interventions: Other: Water exchange colonoscopy

INTERVENTIONS:
Other: Air colonoscopy — Colonoscopy will be performed with conventional air insufflation during colonoscope insertion.
  Arms: Air colonoscopy
Other: Water exchange colonoscopy — Water exchange method (The air pump was turned off before colonoscopy. During colonoscope insertion, residual air in lumen was suctioned and 37°C water was infused into lumen to obtain lumen visualization) was used in whole or left colon. Air was insufflated until cecum was reached or appendix opening was seen.
  Other Names: Water aided colonoscopy
  Arms: Whole-colon water exchange colonoscopy; left-colon water exchange colonoscopy

SUMMARY:
In most of situation, left colon (especially SD junction) is considered the most difficult part of colonoscopy, where endoscopist may encounter difficulty for scope insertion and patients may feel pain or uncomfortable. It is suggested more than half of the whole time for scope insertion should be used in left colon. Many methods, such as water immersion, abdominal palpation, have been used to facilitate insertion in left colon.

Colonoscopy with whole-colon water exchange method has been shown to be useful for reducing medication used, pain experienced during colonoscopy, increasing the success rate of cecum intubation and adenoma detection rate in sedated and unsedated patients undergoing screening colonoscopy. Exchange of water during scope insertion minimizes loop formation and prevents lengthening and distension of the colon during colonoscopy. This will facilitate the colonoscopy in average or difficult colonoscopy. However, it is not known whether the benefits of water exchange method of colonoscopy was mainly due to its effect on the left colon.

We hypothesized that left-colon water exchange colonoscopy (LWE) may have the similar effect regarding the maximal pain score and mean pain score in unsedated patients compared with whole-colon water exchange colonoscopy (WWE). At the mean time, LWE may reduce the insertion time compared with WWE. Here we performed a prospective, randomized controlled study to investigate the efficacies of whole-colon water exchange, left-colon water exchange and air methods of colonoscopy on pain score and insertion time in unsedated outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with unsedated colonoscopy

Exclusion Criteria:

* history of colon resection
* severe colonic stricture or obstructing tumor
* hemodynamic instability
* current pregnancy
* inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cecum intubation time | up to three months
  Insertion time from rectum to reach the cecum.

SECONDARY OUTCOMES:
Pain scores | up to two months
  Pain scores include mean pain score and maximal pain score.
  Mean pain score: mean value of patient reported pain score during the insertion phase in three part of colon by using the visual analog pain scale (0=no pain and 10=most severe pain imaginable).
  Maximal pain score: maximal value of patient reported pain score during the insertion phase in three part of colon by using the visual analog pain scale (0=no pain and 10=most severe pain imaginable).
Polyp detection rate | up to six months
  The proportion of subjects with at least one polyp.
Total procedure time | up to two months
  Total time of colonoscopic procedure.
Cecal intubation rate | up to two months
  Percentage of successful colonoscopy (insertion of colonoscope into cecum).
Withdrawal time | up to two month
  Withdrawal time is defined as the time from withdrawal of the colonoscope from the cecum to anal verge. (This time is measured independent of any therapeutic maneuvers, such as biopsy or polypectomy.)
Patients willingness to repeat colonoscopy using same method | up to two month
  When after the colonoscopic examination, patients were asked if they have willingness to repeat the colonoscopy using same method.
Procedure difficulty evaluated by endoscopist | up to two month
  When after the colonoscopy, endoscopist were asked to score on the difficulty of the colonoscopic procedure.
  0-very easy, 10-very difficult

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, M.D., Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi’an, Shanxi, China

REFERENCES:
- [Derived] Wang X, Luo H, Xiang Y, Leung FW, Wang L, Zhang L, Liu Z, Wu K, Fan D, Pan Y, Guo X. Left-colon water exchange preserves the benefits of whole colon water exchange at reduced cecal intubation time conferring significant advantage in diagnostic colonoscopy - a prospective, randomized controlled trial. Scand J Gastroenterol. 2015 Jul;50(7):916-23. doi: 10.3109/00365521.2015.1010569. Epub 2015 Feb 1. PMID 25639787